CLINICAL TRIAL: NCT04309396
Title: Clinical Utility of Handheld Hydrogen Breathalyzer in Identification of Non-immune Mediated Food Sensitivities (AIRE Study)
Brief Title: Clinical Utility of Handheld Hydrogen Breathalyzer in Identification of Food Sensitivities (AIRE Study)
Acronym: AIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: FoodMarble (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00204104
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: SIBO; Small Bowel Bacterial Overgrowth Syndrome
Keywords: SIBO

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Breath analyzer (Experimental): Candidates who, after the screening period are eligible to receive the AIRE device.
  Interventions: Device: Hydrogen content recording

INTERVENTIONS:
Device: Hydrogen content recording — Eligible participants will eat participants' normal, typical diets during the first week of the study. Participants will use the AIRE machine to measure exhaled H2 content before and after two meals each day - the first meal of the day and the last meal of the day. Participants will breathe into the AIRE machine before eating to obtain a baseline value. Once participants have finished eating, participants will breathe into the AIRE machine 30 minutes, 60 minutes, and 90 minutes postprandially. The participants will record participants' food intake and symptoms directly into participants' smartphone via an app that comes with the AIRE device.

SUMMARY:
Small intestinal bacterial overgrowth (SIBO) is defined as a condition in which an abnormally high amount of coliform bacteria is present in the small bowel and results in premature anaerobic fermentation of carbohydrates before reaching the colon. Commonly recognized causes include gastric achlorhydria, post-surgical bowel stasis, gastrocolic/coloenteric fistulas, and motility disorders leading to bowel stasis.. The current "gold standard" for the diagnosis of SIBO, is a breath test that measures the concentration of hydrogen in response to lactulose, a carbohydrate that is only metabolized by bacteria. However, its accuracy is only about 50% and therefore it is not a very useful test, leading most physicians to treat these patients empirically based on clinical suspicion alone. The purpose of this study is to evaluate the clinical utility of a portable medical device called AIRE, an over-the-counter, commercially available handheld breath analyzer that measures exhaled hydrogen content.

DETAILED DESCRIPTION:
Small intestinal bacterial overgrowth (SIBO) is defined as a condition in which an abnormally high amount of coliform bacteria is present in the small bowel and results in premature anaerobic fermentation of carbohydrates before reaching the colon. Commonly recognized causes include gastric achlorhydria (i.e. due to longstanding proton pump inhibitor (PPI) use), post-surgical bowel stasis, and gastrointestinal motility disorders leading to bowel stasis. Although SIBO is commonly suspected, a major limitation in the field is the lack of a highly accurate test for SIBO. The current gold standard relies on the demonstration of an early rise in breath hydrogen concentration in response to an orally ingested carbohydrate (commonly, lactulose) but its accuracy is about 50%. This may be because it is a one-time snapshot with an artificial substrate. Further, it has to be performed in a clinic, takes up to 5 hours and is relatively expensive. The purpose of this study is to evaluate the clinical utility of a portable medical device called AIRE, which is a validated and commercially available handheld breathalyzer that measures hydrogen content in the breath and connects via Bluetooth to an associated smartphone application to provide immediate results and visual feedback after use.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older)
* Chronic (>3 months) GI symptoms such as nausea, bloating, distention, altered bowel movements, weight loss or abdominal pain with no structural cause other than scleroderma.
* Clinical diagnosis of SIBO by patient's gastroenterologist with plans to obtain a lactulose hydrogen breath test.
* Ability to tolerate oral intake.
* Ability to undergo the LHBT.
* Access to a smartphone with Bluetooth capability

Exclusion Criteria:

* History of current or recent antibiotic use within the last 30 days
* History of inflammatory bowel disease
* Currently following a restrictive diet (for example low Fermentable Oligo-, Di-, Mono-saccharides And Polyols (FODMAP) diet)
* Unable to tolerate oral intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Treisman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 participants were enrolled, however 2 patients withdrew for the study before randomization.
Period: Overall Study
Arm/Group | Breath Analyzer
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Breath Analyzer
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hydrogen Content in Parts Per Million (Ppm)
Description: Exhaled hydrogen (H2) content as measured over a 1-week period by AIRE on the patient's usual diet at home. Mean of one week readings is reported.
Time Frame: Up to 1 week
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Breath Analyzer
Number analyzed (Participants) | 43
ppm | 3.5 (0.7)

2. Primary Outcome: Hydrogen Content in Parts Per Million (Ppm)
Description: For participants who have a positive LHBT test at baseline, antibiotics are prescribed as part of standard of care. These participants will have a repeat AIRE test at 2 weeks post antibiotic treatment.
Time Frame: 2 weeks after antibiotic treatment for positive LHBT
Population: Only participants with positive LHBT test at baseline were analyzed.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Breath Analyzer
Number analyzed (Participants) | 39
ppm | 10.7 (1.1)

3. Primary Outcome: Hydrogen Content in Parts Per Million (Ppm)
Description: For participants who have a negative LHBT test at baseline, a repeat AIRE test is done at 1 month after baseline test.
Time Frame: One month after negative LHBT
Population: Only Participants who had a negative LHBT test at baseline were analyzed
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Breath Analyzer
Number analyzed (Participants) | 4
ppm | 8.5 (3.1)

ADVERSE EVENTS:
Time Frame: Up to 1 month of study participation
Arm/Group | Breath Analyzer
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT04309396/Prot_SAP_ICF_000.pdf